CLINICAL TRIAL: NCT04749680
Title: Comparison of Efficacy and Tolerability of APD Treatment With Different PD Cyclers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry); James Motta, Clinical Research Associate (CRA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PD-Silencia-01-CL
Record Dates: First submitted 2021-01-26; First posted 2021-02-11 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Peritoneal dialysis; Automated peritoneal dialysis (APD); PD cyler; Renal replacement therapy
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, multicentre, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peritoneal dialysis PD (Experimental): Treatment for 2 weeks either with the comparators PD-Night or Homechoice PD cycler depending on the previous treatment (clinical phase I). At the end of these 2 treatment weeks and a subsequent training phase which up to 3 weeks, treatment with the Silencia PD cycler for 2 further weeks (clinical phase II).
  Interventions: Device: PD cycler Silencia

INTERVENTIONS:
Device: PD cycler Silencia — Treatment for 2 weeks either with PD-Night or Homechoice PD cycler (Comparators) depending on the previous Treatment ((clinical phase I). At the end of these 2 treatment weeks and a subsequent training phase which up to 3 weeks, treatment with the Silencia PD cycler for 2 further weeks (clinical phase II).

SUMMARY:
The study has been designed in order to investigate the performance and safety of the new Silencia PD cycler including the Silencia tubing system in comparison to the PD-Night and Homechoice PD cycler which are both well-established PD cyclers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorised physician
* CKD patients being treated with APD for at least 3 months
* Minimum age of 18 years
* Body weight ≥ 40 kg
* Fluid status regularly monitored with Body Composition Monitor (BCM)
* Patients planned to change to the Silencia PD cycler
* Proper functioning catheter
* Intraperitoneal Pressure (IPP) ≤ 18 cm H2O for the maximum of TAVO parameter "permitted patient volume"
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Patients who have any condition prohibiting the use of BCM, like patients with major amputations (e.g. lower leg)
* Patients receiving polyglucose containing PD solution
* Any conditions which could interfere with the patient's ability to comply with the study
* Patients who suffer from peritonitis/exit site infection during the last 4 weeks
* Women of childbearing age without effective means of contraception, pregnancy (pregnancy test will be conducted at start and end of study) or lactation period
* Life expectancy < 3 months
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Total Kt/V urea | at the beginning and end of clinical phase 1 and 2 (each clinical phase is 14 days)
  Measurement of solute removal during peritoneal dialysis focuses on urea
Achieving Kt/Vurea ≥ 1.7 | at the beginning and end of clinical phase 1 and 2 (each clinical phase is 14 days)
  Measurement of solute removal during peritoneal dialysis focuses on urea
Mean daily ultrafiltration (UF) | at the beginning and end of clinical phase 1 and 2 (each clinical phase is 14 days)
  Daily ultrafiltration reached by the Patient with APD

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Machuca, Dr, Principal Investigator — Fresenius Medical Care Chile S.A.
Locations (4):
- Chile (4):
  - Nephocare La Serena, La Serena
  - Nephocare Independencia, Santiago
  - Nephocare Providencia, Santiago
  - Nephocare San Bernardo, Santiago

IPD SHARING:
Plan to Share IPD: No